CLINICAL TRIAL: NCT04199481
Title: A Prospective, Observational, Monocentre 5-year Follow-up Clinical Trial on a Historical Consecutive Cohort of Unicompartmental Knee Arthroplasty Patients Treated With the Mobile Bearing Unicondylar Knee Prosthesis Univation XM
Brief Title: Univation XM France
Status: Withdrawn | Type: Observational
Why Stopped: Study stopped due to product discontinuation by manufacturer
Sponsor: Aesculap AG (Industry)
Collaborators: B. Braun Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1822
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis, Knee; Osteoarthrosis of Knee; Arthritis Knee; Unicompartmental Knee Arthroplasty
Keywords: unicompartmental knee arthroplasty; retrospective study; Knee Society Score
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The study is set up due to regulatory purposes and to collect routine clinical data of the mobile-bearing implant univation XM. The study is designed as a prospective follow-up study with a historic patient cohort who have been treated with the product under investigation two years ago. This design is selected to quicker realize follow-up data as patients have already been treated in the past.

As the mobile version of the implant is not widely used, the study will be set up as a monocentric study in France. The clinical hypothesis of the study is that patients who are treated with the product under investigation have a similar outcome and survival rate in comparison to other established unicondylar knee systems on the market. Comparison for the later evaluation will be taken out of recent orthopaedic registries.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received a primary mobile bearing UKA at the study site between January 2017 and December 2018 using the product under investigation
* Patient's written consent and willingness to participate at the clinical study and the follow-up examinations

Exclusion Criteria:

* Pregnancy
* Patient Age <18 years at the time of the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of the Implant | 5 years after surgery
  Revision-free survival rate after 5 years according to Kaplan-Meier

SECONDARY OUTCOMES:
Development of Knee joint function | in the postoperative course, up to 5 years after surgery
  Postoperative Development of knee joint function measured with the Knee Society Score (KSS). The KSS is composed of two subgroups "Knee Score" and "Function Score"; both parts have a maximum score of 100, where higher values represent better results.
Development of Oxford Knee Score | in the postoperative course, up to 5 years after surgery
  A patient-reported outcome instrument which contains 12 questions on activities of daily living that assess function and residual pain in patients undergoing total knee replacement (TKR) arthroplasty. Oxford Knee Score has a maximum of 48 points indicating satisfactory knee function
Intraoperative/surgery Data | intraoperative
  Surgical and intraoperative data collected will include the date and duration of the surgery, selected implants and sizes, blood loss and implant descriptions. Surgical duration is to be measured from the time of incision to the time of skin closure, skin-to-skin. All potential Adverse Events will be collected during the surgical procedure and/or from the surgical record and will be documented on the intra-operative Evaluation Form.
Radiographic evaluation | in the postoperative course, up to 5 years after surgery
  The outcome and function of a knee prosthesis is influenced by the postoperative alignment of the leg and the orientation in reference to the axis. Incorrect positioning can lead to an increased implant wear and functional limitations; The aim of a postoperative alignment within 3° varus to 3° valgus will be assessed using long leg x-rays up to 5 years after surgery
Rate of Serious Adverse Events | in the postoperative course, up to 5 years after surgery
  As part of the follow-up examination, any upcoming (serious) adverse device events or effects related or not related to the product under investigation, will be documented in the dedicated Case Report Forms. Recorded complications will be categorized and analyzed in order to assess the safety of the univation XM prosthesis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Hopital Hautepierre, Strasbourg, France